CLINICAL TRIAL: NCT04091776
Title: Sensitivity of CT-scan as a Predictor of Fixation Failure in Per-trochanteric Fractures
Brief Title: CT Scan in Per-trochanteric Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Saeed Younis (Other)
Responsible Party: Sponsor-Investigator, Ahmed Saeed Younis, Registrar of orthopaedic surgery, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12376593
Record Dates: First submitted 2019-09-02; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Hip Fractures; Sensitivity; Computed Tomography Scan
MeSH Terms: conditions — Hip Fractures; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT scan — 1. Quantitative CT scan to measure localized osteoporosis and detection of cortices comminution.
  2. Blinded surgeon decision as regard to replace or to fix using DHS or PFN (depending on x-rays data only).
  3. Pathological assessment of osteoporosis in retrieved bone in patients whom hip replacement was decided.
  4. Assessment of fixation failure in fixed fractures if occurred.
  5. Fixation failure is defined as:
  5.1. Lag cut through 5.2. Lag cutout 5.3. Z-effect (lag penetration) 5.4. Non-union (within 6 months) 5.5. Loss of reduction with progressive varus deformity 5.6. Femoral fracture 5.7. Intra-operative fracture of lateral wall or anterior cortex

SUMMARY:
To assess the importance Of Ct scan in the prediction of fixation failure of per-trochanteric fractures

DETAILED DESCRIPTION:
Recently, epidemiological studies had shown an increase in hip fractures with aging of the population. Osteoporosis had been defined by a mean of -2.5 SD upon DEXA scan, which is not a practical tool to use in patients with recent hip fractures until management of such fractures either with fixation or replacement. Also it have been found that assessment of osteoporosis using the Singh index is not a reliable method for osteoporosis diagnosis .

Osteoporosis may affect the decision making for dealing with per-trochanteric fractures as some surgeons prefer to do hip replacement for fear of fixation failure, while others still convinced that fixation with good reduction and appropriate placement of lag screw within a TAD less than 25mm is the best even with unstable types specially after the progress in proximal femoral nails .

CT scan can be used for osteoporosis measurement. Even it can detect stress fractures that are not dRecently, epidemiological studies had shown an increase in hip fractures with aging of the population . Osteoporosis had been defined by a mean of -2.5 SD upon DEXA scan , which is not a practical tool to use in patients with recent hip fractures until management of such fractures either with fixation or replacement. Also it have been found that assessment of osteoporosis using the Singh index is not a reliable method for osteoporosis diagnosis .

Osteoporosis may affect the decision making for dealing with per-trochanteric fractures as some surgeons prefer to do hip replacement for fear of fixation failure, while others still convinced that fixation with good reduction and appropriate placement of lag screw within a TAD less than 25mm is the best even with unstable types specially after the progress in proximal femoral nails .

CT scan can be used for osteoporosis measurement. Even it can detect stress fractures that are not diagnosed using DEXA scan. It can be used to assess BMD in specific regions like spine or hip in a quantitative manner that can be compared to the T score used with DEXA scan . Again It can assess the presence of comminution in the anterior and posterior cortices that might not be easy with x-rays. The thickness of the lateral wall can be better measured through CT scan which is a critical measure while deciding to fix trochanteric fractures using whether DHS or PFN .

The purpose of this prospective clinical cohort study is to assess the sensitivity of CT scan for localized osteoporosis detection that can be used in patients with hip fracture and detection of comminution and thin trochanteric lateral wall that might not be accessible with x-rays. And whether these independent factors could predict the fixation failure iagnosed using DEXA scan. It can be used to assess BMD in specific regions like spine or hip in a quantitative manner that can be compared to the T score used with DEXA scan . Again It can assess the presence of comminution in the anterior and posterior cortices that might not be easy with x-rays. The thickness of the lateral wall can be better measured through CT scan which is a critical measure while deciding to fix trochanteric fractures using whether DHS or PFN .

The purpose of this prospective clinical cohort study is to assess the sensitivity of CT scan for localized osteoporosis detection that can be used in patients with hip fracture and detection of comminution and thin trochanteric lateral wall that might not be accessible with x-rays. And whether these independent factors could predict the fixation failure

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Pertrochanteric fracture requiring surgical treatment
* Ability to understand the content of the patient information
* Informed Consent Form (ICF)
* Willingness and ability to participate in the study
* Signed and dated IRB/ ECs-approved written informed Consent
* Mental capacity to comply with post-operative regimen, evaluation and data collection
* Ability to attend post-operative follow up visits

Exclusion Criteria:

* Known pathological fractures otherwise osteoporosis
* Prisoner
* Unable / unwilling to provide consent

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
CT scan lateral wall integrity (thickness measurement) | one year
  in millimeters

SECONDARY OUTCOMES:
Patients' history (e.g. Charlson comorbidity index) and demographics | one year
  patients, demographics
CT scan detected comminution | one year
QCT measurement of BMD | one year
  QCT radiological measure of bone mineral density
Fixation quality | one year
  expert opinion in fixation quality
Functional and patient reported outcome scores | one year
  e.g Harris hip score HHS
Postoperative complications | one year
  e.g. lag cut out, breal through

CONTACTS AND LOCATIONS:
Overall Officials: Radwan Metwally, Dr., Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No